CLINICAL TRIAL: NCT00564603
Title: Intravenous Continuous Infusion of Dexamethasone Plus Tramadol Combined With Standard Morphine Patient-Controlled Analgesia After Total Abdominal Hysterectomy
Brief Title: Continuous Infusion of Dexamethasone Plus Tramadol Adjunct to Morphine PCA After Abdominal Hysterectomy
Acronym: DTMPCA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Collaborators: HRSA/Maternal and Child Health Bureau (U.S. Federal Agency)
Responsible Party: XiaoFeng Shen, Nanjing Maternal and Child Health Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NMU-2579-5FW; 06NMUZ028
Record Dates: First submitted 2007-11-26; First posted 2007-11-28 (Estimated); Last update posted 2008-04-21 (Estimated); Status verified 2008-04

CONDITIONS: Postoperative Pain; Post Operative Analgesia; Patient-Controlled Analgesia; Abdominal Surgeries
Keywords: Glucocorticoid; Opioids; Balanced analgesia
MeSH Terms: conditions — Pain, Postoperative | interventions — dexamethasone 21-phosphate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): Saline with same volume added to tramadol infusion combined with morphine PCA.
  Interventions: Other: 0.9% Saline
- 2 (Active Comparator): Dexamethasone 10mg in 2mL added to tramadol infusion adjunct to morphine PCA.
  Interventions: Drug: Dexamethasone Sodium Phosphate Injection

INTERVENTIONS:
Drug: Dexamethasone Sodium Phosphate Injection — Dexamethasone, 10mg, continuously infused up to 48h after surgeries.
  Arms: 2
Other: 0.9% Saline — Saline, in same volume of 2mL
  Arms: 1

SUMMARY:
Dexamethasone has been recognized as an antiemetic agent after surgeries, and the combination of dexamethasone and tramadol remained stable in solution up to 5 days. In addition, i.v. basal infusion of tramadol is a certified technique in postoperative pain management. We purposed that combined administration of dexamethasone and tramadol adjunct to i.v. morphine is an effective way in treating postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status I-II
2. Chinese
3. 19-64yr
4. Uterus myoma

Exclusion Criteria:

1. Allergy to opioids, a history of the use of centrally-acting drugs of any sort, chronic pain and psychiatric diseases records.
2. Participants younger than 18yr，older than 65yr or pregnancy was eliminated.
3. Due to the significant changes in vital signs might affect cognition of pain and that of sensation, over 20% variation of these records from the baselines or below 92% of SpO2 under 20-40% nasal tube oxygen at any time should be excluded from the study.
4. Those who were not willing to or could not finish the whole study at any time.
5. Any patient who exhibited a combative or incoherent state of PCA analgesia would be excluded from the study.

Ages: 19 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2007-08; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) of pain | 0-48h after surgeries

SECONDARY OUTCOMES:
First requirement of morphine; Total morphine consumption; VAS sedation; VAS satisfaction; Side effects; Overall conditions of patients; | 0-48h after surgeries

CONTACTS AND LOCATIONS:
Overall Officials: XiaoFeng Shen, MD, Study Director — Nanjing Medical University
Locations (1):
- Nanjing Maternal and Child Care Hospital, Nanjing, Jiangsu, China